CLINICAL TRIAL: NCT03473080
Title: Feasibility of a Therapist and Parent Guided eHealth Intervention for Obsessive Compulsive Disorder in Youth With Autism Spectrum Disorder
Brief Title: An eHealth Intervention for Obsessive Compulsive Disorder in Youth With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Fabian Lenhard, PhD, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIP ASD/OCD pilot
Record Dates: First submitted 2018-02-16; First posted 2018-03-22 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; ASD; Obsessive Compulsive Disorder; Autism Spectrum Disorder; ICBT; eHealth; Internet; CBT; Pediatric; Adolescents; Children; Internet-delivered
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet CBT (Other): Participants and their parents receive 16 weeks of internet-delivered cognitive behavior therapy (CBT) with psychologist support.
  Interventions: Behavioral: Internet CBT

INTERVENTIONS:
Behavioral: Internet CBT — The treatment consists of a standard cognitive behavior therapy for OCD with additional treatment components to make the treatment better suited for children and adolescents with Autism Spectrum Disorder.
  Other Names: ICBT; Internet-delivered Cognitive Behavior Therapy

SUMMARY:
This study is a feasibility study of Internet-delivered CBT for OCD in children and adolescents (7-17 years) with comorbid Autism Spectrum Disorder.

DETAILED DESCRIPTION:
The main objectives of this study is to evaluate the feasibility, acceptability and preliminary efficacy of internet-delivered Cognitive Behavioral Therapy (ICBT) for Obsessive Compulsive Disorder (OCD) in children and adolescents (7-17 years) with Autism Spectrum Disorders (ASD). The study will an open trial with-in group mean comparison design (n=18). The treatment is delivered over 16 weeks. Study participants will be followed up at 3 (primary endpoint), 6 and 12 months after completed treatment. ICBT is expected to decrease OCD-symptoms.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of OCD according to DSM-5
* a diagnosis of autism according to DSM-IV or DSM-5, confirmed with the Autism Diagnostic Interview- Revised or Autism Diagnostic Observation Schedule version 1 or 2 and by medical records
* a total score of ≥ 16 on the Children's Yale-Brown Obsessive-Compulsive Scale
* age between 7 and 17 years
* ability to read and write Swedish
* access to the internet
* a parent that is able to co-participate in the treatment
* participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment

Exclusion Criteria:

* a diagnosis of psychosis, bipolar disorder, severe eating disorder or intellectual disabilities
* comorbid hoarding disorder or OCD with hoarding as a principal symptom.
* suicidal ideation
* subject not able to read or understand the basics of the ICBT material
* completed CBT for OCD within last 12 months (defined as at least 5 sessions of CBT including exposure and response prevention)
* ongoing psychological treatment for OCD or any anxiety disorder
* OCD treatment is not an immediate priority

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale | Baseline, 16 weeks (= post treatment), 3 months after post treatment, 6 months after post treatment, 12 months after post treatment
  Changein obsessions and compulsions will be measured as the total score on the scale.. Total score ranges from 0 to 40 points, a higher score indicates more severe OCD. The scale is rated by a clinician.

SECONDARY OUTCOMES:
Obsessive-compulsive inventory - child version | Baseline, weekly during treatment, 16 weeks (= post treatment), 3 months after post treatment, 6 months after post treatment, 12 months after post treatment
  Child-rating of OCD symptoms. The total score range is 0-42, a higher score indicates more OCD-symptoms.
Autism spectrum quotient (AQ-10) | Baseline
  Parent-rated, brief screeing for symtoms relating to autism spectrum disorder. Total score ranges from 0-10, a higher score indicating more symtoms.
Education, work and social adjustment scale - child and parent version | Baseline, 16 weeks (= post treatment), 3 months after post treatment, 6 months after post treatment, 12 months after post treatment
  Self-rated and parent-rated. Ranges from 0 to 40 points, a higher score indicating more problems. Measures how much the psychiatric problems affect daily life in different areas.
Family accommodation scale for obsessive-compulsive disorder | Baseline, 16 weeks (= post treatment), 3 months after post treatment, 6 months after post treatment, 12 months after post treatment
  Parent-rated scale, total score ranges from 0 to 76, a higher score indicates more family accommodation to the child's OCD.
Mood and Feeling Questionnaire - child and parent version | Baseline, 16 weeks (= post treatment), 3 months after post treatment, 6 months after post treatment, 12 months after post treatment
  Self-rated and parent-rated. Measures depressive symptoms in the child. Total score ranges from 0 to 26, a higher score indicates more depressive symptoms.
Children's Obsessional Compulsive Inventory Revised - parent rated (ChOCI-R-P) | Baseline, weekly during treatment, 16 weeks (= post treatment), 3 months after post treatment, 6 months after post treatment, 12 months after post treatment
  Parent-rated. Consists of 4 Subscales. Obsessive symptoms, Compulsive symtoms, Obsessive impairment and Compulsive impairment. The symptom subscales range from 10 to 30 points, a higher score indicating more symptomology. These subscales are added to get a total score for OCD-symptoms. The score of each impairment subscales ranges from 0 to 24, a higher score indicating more impairment. The score of the impairment subscales are added to get a total score of impairment. The symptom subscales will only be administered at baseline. The impairment subscales will be administered at all assessment points.
Mini International Neuropsychiatric Interview for Children and Adolescents | Baseline
  Clinician-rated, a semi-structured interview to asses psychiatric problems in children. Results will be presented as co-morbid psychiatric diagnoses.
Children's global assessment scale | Baseline, 16 weeks (= post treatment), 3 months after post treatment, 6 months after post treatment, 12 months after post treatment
  Clinician-rated, measures the childs global psychiatric functioning. Total score ranges from 0-100, a lower score indicates lower functioning.
Children's Assessment Scale for Developmental Disabilities | Baseline
  Clinician-rated. measures the childs global functioning with respect to developmental disabilities. Total score ranges from 0 to 100, a lower score indicates lower functioning.
Clinical global impression - severity | Baseline, 16 weeks (= post treatment), 3 months after post treatment, 6 months after post treatment, 12 months after post treatment
  Clinician-rated level of psychiatric severity, the score ranges from 1 to 7, a lower score indicates less severity. In this study the measure will only refer to level of OCD.
Clinical global impression - improvement | 16 weeks (= post treatment), 3 months after post treatment, 6 months after post treatment, 12 months after post treatment
  Clinician-rated level of psychiatric improvement, the score ranges from 1 to 7, a lower score indicates more improvement. In this study the measure will only refer to level of OCD.
internet intervention Patient Adherence Scale | 8 weeks, 16 weeks
  Clinician-rated, measures the patients adherence to treatment. The scale consist of 5 items measuring 1. If the patient is in phase with treatment, 2, level of engagement in treatment 3, level of communication with the clinician, 4 motivation to change 5, frequency of log-ins to the internet-treatment. Total score ranges from 0 to 20, a higher score indicates more adherence to the treatment.
Client Satisfaction Questionnaire (CSQ-8) | 16 weeks
  Self-rated and parent-rated. Measures level of satisfaction with the treatment. Total score ranges from 8 to 32, higher level indicates higher satisfaction.
Parent strategies | Post-treatment
  A parent-rated questionnaire consisting of 4 items measuring the parents 1, participation in treatment, 2, cooperation with the child during treatment, 3, autonomus support in treatment and 4, directiveness in treatment. The questions are qualitative and results will be presented on an item level
Patient EX/RP Adherence Scale | Weekly for 16 weeks (during treatment)
  Self-rated questionnaire. Consist of 3 items: 1, percentage of attempted exposure exercises, 2, how well exposures were performed and 3, percentatge of respons-prevention during the last week. The answers will be presented on an item level.
Drop-out rate from treatment | at week 16
  Percentage of patients that drop out from ICBT
Completed treatment modules | week 16
  Number of completed treatment modules

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Lenhard, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- BUP OCD and Related Disorders, Stockholm, Sweden